CLINICAL TRIAL: NCT05533463
Title: Phase I Study to Evaluate the Safety ,Tolerability, and Pharmacokinetics of HRS-4642 in Patients With Advanced Solid Tumors Harboring KRAS G12D Mutation
Brief Title: Phase I Study of HRS-4642 in Patients With Advanced Solid Tumors Harboring KRAS G12D Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4642-I-101
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced KRAS G12D Mutant Solid Tumors

STUDY DESIGN:
Intervention Model Description: Single arm study of HRS-4642
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-4642 (Experimental): In Dose Escalation:
  HRS-4642 will be injected QW. Six dose levels are preset.
  In Dose Expansion:
  1 to 2 dose cohorts will be selected for dose expansion stage.
  In Indication Expansion:
  Enrollment into the dose expansion cohorts may be from any eligible solid tumor type.
  Interventions: Drug: HRS-4642

INTERVENTIONS:
Drug: HRS-4642 — HRS-4642 will be administrated per dose level in which the patients are assigned.

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of HRS-4642 in patients with advanced solid tumors harboring KRAS G12D mutation.To estimate the maximum tolerated dose (MTD) and/or a biologically active dose (eg, recommended phase 2 dose [RP2D]) within investigated subject population groups

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old.
3. Histologically confirmed diagnosis of advanced solid tumor harbouring with KRAS G12D mutation
4. ECOG performance status of 0-1.
5. With a life expectancy of ≥3 months.
6. Have at least one measurable lesion.
7. Adequate laboratory parameters during the screening period

Exclusion Criteria:

1. Previously received KRAS G12D inhibitors
2. Priot radiotherapy within 28 days for non-thoracic radiation
3. Prior anti-tumor chemotherapy (< 6 weeks if chemotherapy including nitrosoureas or mitomycin) within 4 weeks before the study drug administration
4. Any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or inclusion/exclusion criteria level (The investigators determined that safe and controllable toxicity was excluded, such as alopecia and ≤ grade 2 peripheral neuropathy ).
5. Central nervous system (CNS) metastases
6. Major surgical therapy within 28 days prior to the date of signature of informed consent form, or expected major surgery during the study.
7. Known history of hypersensitivity to any components of HRS-4642.
8. Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: adverse events(AEs), serious adverse events（SAEs）. | 24 months
  Assess safety and tolerability of HRS-4642 by way of adverse events (CTCAE v5.0).
Dose Limited Toxicity(DLT) | from day 1 to Day 21
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 Day 1 (C1D1), excluding toxicities clearly related to disease progression or intercurrent illness
Maximum tolerated dose (MTD) | From Day 1 to Day 21
  Incidence and category of dose limiting toxicities (DLTs) during the first 21-day cycle of HRS-4642 treatment.
RP2D | 24 months
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in dose escalation and dose expansion stages.

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | 24months.
Number of subjects with clinically significant changes in ECOG, vital signs and physical examination. | 24months.
Number of subjects with changes on ECG. | 24months.
Efficacy endpoints: Overall response rate (ORR). | 24months.
  Evaluated by RECIST v1.1.
Efficacy endpoints: Duration of response (DoR). | 24 months.
  Evaluated by RECIST v1.1
Efficacy endpoints: Disease control rate (DCR). | 24months.
  Evaluated by RECIST v1.1.
Efficacy endpoints: Progression free survival (DoR). | 24months.
  Evaluated by RECIST v1.1.
Efficacy endpoints: overall survival (OS). | 24minths
  Evaluated by RECIST v1.1
Cmax. | 24 months.
  Maximal plasma concentration.
Tmax. | 24 months
  Time to Cmax.
AUC. | 24 months.
  Area under the plasma concentration-time curve.
t1/2. | 24 months.
  Terminal-phase elimination half-life.
Vz/F. | 24 months.
  Apparent volume of distribution during terminal phase after non-intravenous administration.
CL/F. | 24 months.
  Apparent total clearance of the drug from plasma after oral administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided